CLINICAL TRIAL: NCT07324330
Title: Slowing Cognitive Decline in Alpha-synucleinopathies by Enhancing Physical Activity
Acronym: ALPHA-FIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Collaborators: Radboud University Medical Center (Other); Medical University Innsbruck (Other); IJsfontein B.V., Netherlands (Unknown); Synaptikon GmbH (Unknown); Parkinson Stiftung (Unknown)
Responsible Party: Principal Investigator, Dr. Michael Sommerauer, Senior Consultant Physician, Head of the Sleep Laboratory, University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2025-289-BO; 01EA2501 (Other Grant/Funding Number: Bundesministerium für Forschung, Technologie und Raumfahrt (BMFTR)); 101095426 (Other Grant/Funding Number: Era4Health)
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease; Prodromal Stage; Neurodegenerative Diseases; Basal Ganglia Diseases; Central Nervous System Diseases; Synucleinopathies; Nervous System Diseases; Cerebral Disorder; Brain Diseases; Parkinsonian Disorders
Keywords: intervention; movement; iRBD; prodromal parkinson's; non-pharmacologic; alpha-synucleinopathy; biomarker; cognitive decline; executive function; MRI; lifestyle; prevention; RCT; motor decline; smartphone; smartwatch; accelerometer; scalable; prodromal; PD; Parkinson; Lewy-body; MSA; multiple system atrophy; dementia
MeSH Terms: conditions — Parkinson Disease; Prodromal Symptoms; Neurodegenerative Diseases; Basal Ganglia Diseases; Central Nervous System Diseases; Synucleinopathies; Nervous System Diseases; Brain Diseases; Parkinsonian Disorders; Cognitive Dysfunction; Multiple System Atrophy; Dementia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doubling of baseline step count (Experimental): Large increase in step count and moderate to vigorous physical activity relative to baseline level (+100%).
  Interventions: Behavioral: Increase of physical activity volume and intensity with the use of a motivational smartphone application
- Small increase of baseline step count (Active Comparator): Small increase in step count and moderate to vigorous physical activity relative to baseline level (+10%).
  Interventions: Behavioral: Increase of physical activity volume and intensity with the use of a motivational smartphone application

INTERVENTIONS:
Behavioral: Increase of physical activity volume and intensity with the use of a motivational smartphone application — A motivational smartphone application will be available for all participants using their own smartphone: the Alpha-Fit app, comparable to the SLOW-SPEED app (https://clinicaltrials.gov/study/NCT06993142). The Alpha-Fit app will motivate participants to increase the volume and intensity of their physical activity in daily life over a long period of time (12 months) based on their own baseline levels. Different treatment arms will receive different physical activity goals. The app offers participants feedback and support, that will stimulate them to reach their individual physical activity goal (i.e. incremental relative increase of step count and minutes exerting ≥ 64% of maximum heart rate reflecting moderate-to-vigorous physical activity (MVPA) relative to baseline level).
  Other Names: Motivational movement intervention

SUMMARY:
α-Synucleinopathies, including Parkinson's disease and dementia with Lewy bodies, are the second most common neurodegenerative diseases. In addition to progressive motor deterioration, cognitive decline is a key element of the non-motor symptom complex of these diseases. Isolated rapid eye movement (REM) sleep behavior disorder (iRBD) indicates an early stage of α-synucleinopathies, even before relevant motor or cognitive disorders are present. Therapeutic interventions in individuals with iRBD therefore have great preventive potential. In particular, increasing physical activity could have a relevant effect on neurodegenerative processes, including the preservation of cognitive functions.

The aim of the study is therefore to investigate the effects of increased physical activity in everyday life on cognitive functions in individuals with iRBD. In this randomized, double-blind, actively controlled study, an increase in physical activity will be implemented over a period of one year with the help of a motivational smartphone application. The intervention and control conditions are the same as those used in the Slow-SPEED trials, making the connection between the trials concrete. The primary outcome parameter is the change in cognitive performance in a neuropsychological test battery over one year.

Eighty individuals with iRBD and 50 age- and gender-matched individuals are being recruited at the University Hospital Bonn and the "Deutsches Zentrum für Neurodegenerative Erkrankungen" (DZNE) Bonn (German branch only). In addition to classic neuropsychological tests as the primary endpoint, magnetic resonance imaging (MRI) and blood-based markers of brain aging are being examined as secondary endpoints. This study is in close collaboration with the Slow-SPEED study (https://clinicaltrials.gov/study/NCT06993142). In addition, selected data from three separate trials-Alpha-Fit, Slow-SPEED-NL, and a sister trial in Austria currently in preparation-are planned to be synthesized into a meta-analysis.

DETAILED DESCRIPTION:
α-Synucleinopathies are the second most common group of neurodegenerative diseases after Alzheimer's disease (AD). Their prevalence is expected to increase significantly, with more than 12 million people worldwide likely to be affected by 2040. Clinical manifestations include Parkinson's disease (PD) and dementia with Lewy bodies (DLB). These diseases are characterized by neuronal inclusions of α-synuclein aggregates and Lewy bodies, which lead to premature aging of the brain. In addition to motor impairments, cognitive decline is a central element of non-motor symptoms, which not only occurs in DLB but also affects up to 80% of people with PD. Cognitive deficits can often occur in the early stages of the disease and significantly impair social functioning and quality of life. Despite their high prevalence, there are currently only a few therapeutic approaches for treating cognitive impairments in α-synucleinopathies. Therefore, easily accessible, early preventive interventions are crucial to counteract cognitive decline.

Isolated REM sleep behavior disorder (iRBD) is considered an early sign of α-synucleinopathy and can be reliably diagnosed using video polysomnography. Over 90% of individuals with iRBD develop either PD or DLB within 20 years of diagnosis, with an approximately equal distribution between the two entities. It is noteworthy that executive functions can often already be impaired in iRBD, which is associated with an increased risk of early conversion to PD or DLB. Thus, iRBD represents a phase of early neurodegeneration in which there is a high risk of cognitive decline. For this reason, individuals with iRBD are a particularly suitable target group for investigating the effects of lifestyle modifications that could slow the progression of the disease at an early stage.

Increasing physical activity could offer a promising way to slow the progression of neurodegenerative processes in the early stages of α-synucleinopathies. Since motor impairments are a central feature of PD and DLB, many affected individuals-even in the early stages of the disease-do not achieve the recommended level of physical activity. Studies on increasing physical activity have shown that physical training has positive effects on cerebrovascular function and cognitive performance, both in healthy aging and in various neurodegenerative diseases. For α-synucleinopathies in particular, there is evidence from animal models, observational studies, and clinical trials with up to six months of follow-up that physical activity may have disease-modifying effects. A recent meta-analysis in PD found that various interventions to increase physical activity have moderate effects on global cognition and even strong effects on executive functions. Therefore, promoting a more active lifestyle could be a promising strategy to positively influence the early course of α-synucleinopathies. Motivational mobile apps offer a novel way to increase physical activity, as they can be used completely independently, allowing for a high degree of scalability of the intervention.

Derivation of research questions

The following key questions will be addressed in the research project:

* Can the progression of motor and cognitive changes in individuals with iRBD be influenced by increasing physical activity?
* Does this intervention also affect biological and imaging markers of pathological brain aging?
* Does this intervention also have an effect on healthy older people?

ELIGIBILITY:
Inclusion Criteria:

iRBD:

* Age: 50-80 years
* Polysomnographically confirmed diagnosis of iRBD
* Maximum of 120 minutes of sports/outdoor activities per day
* Less than an average of 10,000 steps per day during the 4-week eligibility and baseline phase
* Basic smartphone skills
* Sufficient knowledge of German (native language, C1 or C2)
* Ownership of a suitable smartphone (minimum screen size 4.6 inches, Android version 9 or iOS version 15 or newer)
* Consent to be informed of any additional findings

Healthy controls:

* Age: 50-80 years
* Maximum of 120 minutes of sports/outdoor activities per day
* Less than an average of 10,000 steps per day during the 4-week eligibility and baseline phase
* Basic smartphone skills
* Sufficient knowledge of German (native language, C1 or C2)
* Ownership of a suitable smartphone (minimum screen size 4.6 inches, Android version 9 or iOS version 15 or newer)
* Consent to be informed of any additional findings

Exclusion Criteria:

iRBD:

* Relevant cardiovascular diseases
* Problems with dexterity or cognitive impairments that make it difficult to use a smartphone
* Cognitive impairments that limit the ability to make informed decisions and consent to participate in the study
* Ownership of one of the following devices: Huawei P8 Lite, Huawei P9 Lite, Xiaomi Mi 6, Huawei P20 Lite (FitBit is not compatible)

Healthy controls:

* Relevant cardiovascular diseases
* Problems with dexterity or cognitive impairments that make it difficult to use a smartphone
* Cognitive impairments that limit the ability to make informed decisions and consent to participate in the study
* Ownership of one of the following devices: Huawei P8 Lite, Huawei P9 Lite, Xiaomi Mi 6, Huawei P20 Lite (FitBit is not compatible)
* clinically diagnosed iRBD

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive Performance: Change in mild cognitive impairment (MCI) in PD Level II Criteria | 12 months
  Change in cognitive performance between the start of the study (baseline) and the time after the intervention (after 12 months of intervention), measured as the global mean of the results from a neuropsychological test battery according to MCI in PD Level II criteria.
  Executive functions:
  * semantic word fluency
  * set-shifting abilities
  * inhibition
  * logical thinking
  Visual cognitive abilities:
  * spatial perception
  * working memory performance
  * processing speed
  * attention
  Memory functions:
  * verbal memory
  * visuospatial memory
  Linguistic abilities:
  * naming semantic
  * abstract thinking

SECONDARY OUTCOMES:
Motor functions: Change in Movement Disorder Society-sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) III | 12 months
  Change in score which ranges from 0 to 108. Higher score indicates greater motor impairment.
Motor functions: Change Perdue-Pegboard-Test | 12 months
  Change in score. Higher scores indicates better manual dexterity and hand coordination.
Motor functions: Change in digital testing outcomes | 12 months
  Change in digital testing assessment, funded by the European Research Council (ERC) (https://cordis.europa.eu/project/id/101169580).
Change in body composition | 12 months
  Change in body composition measured through MRI sequences and bio-electric impedance analysis.
Sleep behavior: Change in subjective sleep quality | 12 months
  Change in Pittsburgh Sleep Quality Index (PSQI), with scores between 0 and 21, higher scores indicate worse sleep.
Sleep behavior: Change in Polysomnography (PSG) read-outs | 12 months
  Change in PSG read-outs.
Change in blood-based markers for metabolism. | 12 months
  Change found in biomarkers in plasma, serum and peripheral blood mononuclear cells (PBMCs).
Change in blood-based markers for neurodegeneration. | 12 months
  Change found in biomarkers in plasma, serum and PBMCs
Change in blood-based markers for inflammation. | 12 months
  Change found in biomarkers in plasma, serum and PBMCs
Cognitive performance: Change in performance in digital app | 12 months
  Change in performance in the https://www.neuronation.com/ app. Will be measured in 2-week intervals.
Change in Quantitative MRI Measures of Brain Structure and Function | 12 months
  Change from baseline to 12 months in MRI-derived quantitative measures of brain structure and function, including resting-state functional magnatic resonance imaging (fMRI), T1-weighted structural measures, fluid-attenuated inversion recovery (FLAIR) based measures, quantitative susceptibility mapping (QSM) metrics, and neuromelanin-sensitive MRI signal measures.

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Sommerauer, Dr., Principal Investigator — University Hospital of Bonn
Locations (1):
- University Hospital of Bonn, Bonn, North Rhine West-Falia, Germany

IPD SHARING:
Plan to Share IPD: Yes
We will make relevant anonymised data available in a database.
Supporting Information: Study Protocol
Time Frame: We will make relevant anonymised data available in a database after publication of the main results of our trial.
Access Criteria: Researchers who are interested in re-use of the data are asked to contact the central contact person for permission.

REFERENCES:
- [Background] Litvan I, Goldman JG, Troster AI, Schmand BA, Weintraub D, Petersen RC, Mollenhauer B, Adler CH, Marder K, Williams-Gray CH, Aarsland D, Kulisevsky J, Rodriguez-Oroz MC, Burn DJ, Barker RA, Emre M. Diagnostic criteria for mild cognitive impairment in Parkinson's disease: Movement Disorder Society Task Force guidelines. Mov Disord. 2012 Mar;27(3):349-56. doi: 10.1002/mds.24893. Epub 2012 Jan 24. PMID 22275317
- [Background] Kim R, Lee TL, Lee H, Ko DK, Lee JH, Shin H, Lim D, Jun JS, Byun K, Park K, Jeon B, Kang N. Effects of physical exercise interventions on cognitive function in Parkinson's disease: An updated systematic review and meta-analysis of randomized controlled trials. Parkinsonism Relat Disord. 2023 Dec;117:105908. doi: 10.1016/j.parkreldis.2023.105908. Epub 2023 Oct 26. PMID 37922635
- [Background] Jia RX, Liang JH, Xu Y, Wang YQ. Effects of physical activity and exercise on the cognitive function of patients with Alzheimer disease: a meta-analysis. BMC Geriatr. 2019 Jul 2;19(1):181. doi: 10.1186/s12877-019-1175-2. PMID 31266451
- [Background] Jellinger KA, Korczyn AD. Are dementia with Lewy bodies and Parkinson's disease dementia the same disease? BMC Med. 2018 Mar 6;16(1):34. doi: 10.1186/s12916-018-1016-8. PMID 29510692
- [Background] Janssen Daalen JM, Schootemeijer S, Richard E, Darweesh SKL, Bloem BR. Lifestyle Interventions for the Prevention of Parkinson Disease: A Recipe for Action. Neurology. 2022 Aug 16;99(7 Suppl 1):42-51. doi: 10.1212/WNL.0000000000200787. PMID 35970584
- [Background] Höglinger, G. U. et al. Towards a Biological Definition of Parkinson's Disease. Preprint at https://doi.org/10.20944/preprints202304.0108.v1 (2023).
- [Background] Fang X, Han D, Cheng Q, Zhang P, Zhao C, Min J, Wang F. Association of Levels of Physical Activity With Risk of Parkinson Disease: A Systematic Review and Meta-analysis. JAMA Netw Open. 2018 Sep 7;1(5):e182421. doi: 10.1001/jamanetworkopen.2018.2421. PMID 30646166
- [Background] Dorsey ER, Sherer T, Okun MS, Bloem BR. The Emerging Evidence of the Parkinson Pandemic. J Parkinsons Dis. 2018;8(s1):S3-S8. doi: 10.3233/JPD-181474. PMID 30584159
- [Background] de Vries NM, Darweesh SKL, Bloem BR. Citius, Fortius, Altius-Understanding Which Components Drive Exercise Benefits in Parkinson Disease. JAMA Neurol. 2021 Dec 1;78(12):1443-1445. doi: 10.1001/jamaneurol.2021.3744. No abstract available. PMID 34724528
- [Background] Dauvilliers Y, Schenck CH, Postuma RB, Iranzo A, Luppi PH, Plazzi G, Montplaisir J, Boeve B. REM sleep behaviour disorder. Nat Rev Dis Primers. 2018 Aug 30;4(1):19. doi: 10.1038/s41572-018-0016-5. PMID 30166532
- [Background] Cesari M, Heidbreder A, St Louis EK, Sixel-Doring F, Bliwise DL, Baldelli L, Bes F, Fantini ML, Iranzo A, Knudsen-Heier S, Mayer G, McCarter S, Nepozitek J, Pavlova M, Provini F, Santamaria J, Sunwoo JS, Videnovic A, Hogl B, Jennum P, Christensen JAE, Stefani A. Video-polysomnography procedures for diagnosis of rapid eye movement sleep behavior disorder (RBD) and the identification of its prodromal stages: guidelines from the International RBD Study Group. Sleep. 2022 Mar 14;45(3):zsab257. doi: 10.1093/sleep/zsab257. PMID 34694408
- [Background] Bliss ES, Wong RH, Howe PR, Mills DE. Benefits of exercise training on cerebrovascular and cognitive function in ageing. J Cereb Blood Flow Metab. 2021 Mar;41(3):447-470. doi: 10.1177/0271678X20957807. Epub 2020 Sep 20. PMID 32954902
- [Background] Berg D, Borghammer P, Fereshtehnejad SM, Heinzel S, Horsager J, Schaeffer E, Postuma RB. Prodromal Parkinson disease subtypes - key to understanding heterogeneity. Nat Rev Neurol. 2021 Jun;17(6):349-361. doi: 10.1038/s41582-021-00486-9. Epub 2021 Apr 20. PMID 33879872
- [Background] Barone P, Antonini A, Colosimo C, Marconi R, Morgante L, Avarello TP, Bottacchi E, Cannas A, Ceravolo G, Ceravolo R, Cicarelli G, Gaglio RM, Giglia RM, Iemolo F, Manfredi M, Meco G, Nicoletti A, Pederzoli M, Petrone A, Pisani A, Pontieri FE, Quatrale R, Ramat S, Scala R, Volpe G, Zappulla S, Bentivoglio AR, Stocchi F, Trianni G, Dotto PD; PRIAMO study group. The PRIAMO study: A multicenter assessment of nonmotor symptoms and their impact on quality of life in Parkinson's disease. Mov Disord. 2009 Aug 15;24(11):1641-9. doi: 10.1002/mds.22643. PMID 19514014
- [Background] Aarsland D, Batzu L, Halliday GM, Geurtsen GJ, Ballard C, Ray Chaudhuri K, Weintraub D. Parkinson disease-associated cognitive impairment. Nat Rev Dis Primers. 2021 Jul 1;7(1):47. doi: 10.1038/s41572-021-00280-3. PMID 34210995